CLINICAL TRIAL: NCT04454307
Title: Safety and Efficacy of Tramadol Adjuvant Therapy to Standard Care for COVID-19 Egyptian Patients: A Randomized Double Blind Controlled Clinical Trial
Brief Title: Safety and Efficacy of Tramadol in COVID-19 Egyptian Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Nahla El-Ashmawy, Dean of Faculty of Pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRAM/COVID19
Record Dates: First submitted 2020-06-29; First posted 2020-07-01 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Tramadol

STUDY DESIGN:
Intervention Model Description: A randomized Double Blind Controlled Clinical Trial
Who Masked: Participant, Care Provider
Masking Description: A randomized Double Blind Controlled Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tramadol (Experimental): tramadol 100 mg twice daily for 10 days
  Interventions: Drug: Tramadol
- standard care (Active Comparator): standard care plus (placebo twice daily for 10 days).
  Interventions: Other: Standard care delivered in the isolation hospitals.

INTERVENTIONS:
Drug: Tramadol — tramadol 100 mg twice daily for 10 days
  Other Names: tramal
  Arms: Tramadol
Other: Standard care delivered in the isolation hospitals. — Oxygen ventilation.
  Other Names: nasal oxygen
  Arms: standard care

SUMMARY:
The rationale of the use of tramadol for COVID-19 patients is attributed to its anti-inflammatory, hypocagulatory, antioxidant, cardio-protective, analgesic, antitussive, bactericidal and antidepressant effect.

DETAILED DESCRIPTION:
Background and Rationale:

T cells play a critical role in antiviral immunity, their level was dramatically reduced in COVID-19 patients. There is a negative correlation between T cell numbers and cytokines serum level in COVID-19 patients. In those patients, there is up-regulation of inflammatory cytokines including interleukin (IL)-1, IL-6, tumor necrosis factor (TNF)-α, and interferon γ. This makes the use of tramadol reasonable in such patients because it has anti-inflammatory effect decreasing plasma level of TNF-α after treatment with a dose of 100 mg every 12 hours for 10 days, which may result in a subsequent increase in T cell numbers.

Besides, COVID-19 patients with acute respiratory failure present with severe hypercoagulability due to hyperfibrinogenemia resulting in increased fibrin formation and polymerization that may predispose to thrombosis. It has been reported that tramadol has a hypocoagulable effect in the blood of women with gynecologic malignancies. Consequently, tramadol may be useful for patients who have a tendency toward a hypercoagulable status and thromboembolic complications. Moreover, tramadol could affect hemostatic parameters in favor of bleeding tendency in rats.

On the other hand, the severity and mortality risk of COVID-19 have been associated with the age. This age-related mortality is attributed to the shortage of antioxidant mechanisms and increased oxidative damage. Tramadol increased the antioxidant enzymes superoxide dismutase and glutathione peroxidase while diminished the oxidative stress marker malondialdehyde in testicular ischemia-reperfusion injury in rats. Owing to its antioxidant properties, tramadol could reduce complications in COVID-19 patients.

Moreover, tramadol was reported to significantly lower lactate dehydrogenase (LDH) level and to provide a cardio-protective effect. This property of tramadol seems beneficial since it was found that, about 60% of COVID-19 patients are presented with elevated LDH levels. Tramadol has also antitussive property. Tramadol is a unique analgesic offering moderate, dose-related pain relief through its action at multiple sites. In contrast to pure opioid agonists, it has a low risk of respiratory depression, tolerance, and dependence. Previous studies confirmed that tramadol dependence may occur when it is used daily for more than a few weeks/months.

More interestingly, patients infected with COVID-19 may experience intense emotional and behavioral reactions, such as fear, loneliness, anxiety, insomnia, or anger. These conditions can be especially prevalent in quarantined patients. Tramadol is a centrally acting analgesic drug with a dual mechanism of action: binding to μ-opioid receptors and the inhibition of serotonin and norepinephrine reuptake. Through its ability to inhibit serotonin and norepinephrine reuptake, tramadol may exhibit antidepressant activity. In this context, the analgesic and antidepressant effects of tramadol may favor its use for COVID-19 patients. Tramadol also was found to have dose- and time-dependent bactericidal activity against Escherichia coli, Staphylococcus aureus, Staphylococcus epidermidis, and Pseudomonas aeruginosa pathogens in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed symptomatic COVID-19 patients with mild to moderate respiratory manifestations, adults (18-65 Years old), and both sexes.

Exclusion Criteria:

* Patients with abnormal liver function (ALT, AST), chronic kidney disease or dialysis (CrCl< 30 ml/min)
* Pregnant women or women who are breastfeeding
* Immunocompromised patients taking medication upon screening
* Subjects with comorbid condition like hypertension, cardiovascular disease, diabetes mellites, asthma, COPD, malignancy
* Patients having allergy to Hydroxychloroquine and/or Nitazoxanide
* Patients with contraindication towards the study medication including retinopathy, G6PD deficiency and QT prolongation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Number of COVID-19 PCR negative cases | 10 days
  PCR analysis of nasal swabs from COVID-19 patients

CONTACTS AND LOCATIONS:
Overall Officials: Nahla Elashmawy, PhD, Principal Investigator — Tanta University

IPD SHARING:
Plan to Share IPD: No